CLINICAL TRIAL: NCT04418427
Title: A Phase 2, Multi-Center, Randomized, Double-Masked, Active Controlled Study of ADVM-022 (AAV.7m8-aflibercept) in Subjects With Diabetic Macular Edema [INFINITY]
Brief Title: ADVM-022 Intravitreal Gene Therapy for DME
Acronym: INFINITY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Adverum Biotechnologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADVM-022-04
Record Dates: First submitted 2020-05-28; First posted 2020-06-05 (Actual); Results first posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Macular Edema; Diabetic Retinopathy
Keywords: ADVM-022; ADVM-022-04; AAV.7m8; Anti-VEGF therapy; Blindness; INFINITY; Gene therapy; Aflibercept (Eylea); Retinal Diseases; Eye Diseases; AAV Vector; Adverum; DME; Diabetic macular edema; Diabetic eye disease; Diabetic retinopathy; DR; AAV.7m8-aflibercept; Ixoberogene soroparvovec; Ixo-vec
MeSH Terms: conditions — Diabetic Retinopathy; Blindness; Retinal Diseases; Eye Diseases | interventions — aflibercept

STUDY DESIGN:
Masking Description: From May 2020 through April 2021: Double-masked study - participants, outcomes assessors and the designated masked study personnel were to have been masked to subject's treatment assignment throughout the study. There must have been a minimum of two physicians per site to fulfill the masking requirements of the study. A masked and unmasked investigator were required to be present for administration of the preceding dose of aflibercept or sham and following dose of ADVM-022 or sham visits, thereafter only the masked investigator was required to be present.
  Starting April 2021: Open label study - study was unmasked for enhanced safety monitoring.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1 (Experimental): 6E11 vg/eye ADVM-022 +/- aflibercept 2mg IVT
  Interventions: Biological: 6E11 vg/eye of ADVM-022; Biological: Aflibercept
- 2 (Experimental): 2E11 vg/eye ADVM-022 +/- aflibercept 2mg IVT
  Interventions: Biological: 2E11 vg/eye of ADVM-022; Biological: Aflibercept
- 3 (Active Comparator): Aflibercept 2mg IVT
  Interventions: Biological: Aflibercept

INTERVENTIONS:
Biological: 6E11 vg/eye of ADVM-022 — ADVM-022 (AAV.7m8-aflibercept) is a recombinant, replication-incompetent adeno-associated virus (AAV.7m8) gene therapy vector carrying a coding sequence for aflibercept
  Other Names: AAV.7m8-aflibercept
  Arms: 1
Biological: 2E11 vg/eye of ADVM-022 — ADVM-022 (AAV.7m8-aflibercept) is a recombinant, replication-incompetent adeno-associated virus (AAV.7m8) gene therapy vector carrying a coding sequence for aflibercept
  Other Names: AAV.7m8-aflibercept
  Arms: 2
Biological: Aflibercept — Commercially available Active Comparator
  Other Names: Eylea

SUMMARY:
A Phase 2, Multi-Center, Randomized, Double-Masked*, Active Controlled Study of ADVM-022 (AAV.7m8-aflibercept) in Subjects with Diabetic Macular Edema [INFINITY]

DETAILED DESCRIPTION:
ADVM-022 (also known as Ixo-vec and AAV.7m8-aflibercept) is an investigational gene therapy product developed for the treatment of serious retinal vascular diseases including Diabetic Macular Edema (DME), a vision-threatening complication of diabetic retinopathy. DME can affect up to 10% of individuals with both type 1 and type 2 diabetes mellitus. Current therapies for treating DME include anti-vascular endothelial growth factor (anti-VEGF) agents that require frequent and long-term intravitreal (IVT) injections to achieve and maintain efficacy. ADVM-022 is intended provide sustained intraocular expression of aflibercept from a single IVT injection to potentially reduce the current treatment burden and prevent disease progression and vision loss due to undertreatment.

This Phase 2, randomized, controlled study (INFINITY) enrolled 36 eligible participants with DME. The participants were randomized to receive one of the two dose levels of ADVM-022 or assigned to the control arm to receive a sham ocular injection with a preceding aflibercept injection. Participants randomized to the ADVM-022 arms were assigned to receive a preceding aflibercept or sham ocular injection. All participants were monitored regularly for disease activity and may have received supplemental aflibercept based on predefined retreatment criteria. All participants were to be followed over a 96- week follow-up period.

To enhance safety monitoring for participants in this study, the sponsor unmasked treatment assignment (in April 2021) due to the occurrence of a suspected unexpected serious adverse reaction (SUSAR) which occurred early in the study in the high dose (ADVM-022 6E11 vg/eye) arm. Interpretation of the results of this study should consider the potential confounding nature of this unmasking in the context of the observed dose-limiting events and the associated additional use of topical/intravitreal/systemic steroids, particularly in the high dose ADVM-022 arm.

In this study ADVM-022 (Ixo-vec) demonstrated improved efficacy across endpoints, reducing the need for supplemental aflibercept in DME management and demonstrating a clinically meaningful delay in DME worsening and improved outcomes across multiple endpoints compared to the control arm (sham + Aflibercept). However, the benefit of the ADVM-022 6E11 vg/eye dose was affected by dose-limiting toxicities in some participants. In terms of safety outcomes, the most common ADVM-022-related adverse events were mild-to-moderate intraocular inflammation, a known and expected side effect of ocular gene therapy, which was generally responsive to corticosteroid eye drops. No Ixo-vec-related events were reported in the fellow eye or systemically, indicating no off-target effects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Type 1 or Type 2 diabetes mellitus
* Willing and able to provide informed consent
* Vision impairment due to center involving diabetic macular edema

Exclusion Criteria:

* Uncontrolled diabetes defined as HbA1C >10%, or history of diabetic ketoacidosis within 3 months prior to randomization; or subjects who, within the last 3 months, initiated intensive insulin treatment (a pump or multiple daily injection) or plan to do so in the next 3 months.
* Acute coronary syndrome, myocardial infarction or coronary artery revascularization, CVA, TIA in the last 6 months
* Uncontrolled hypertension defined as average SBP ≥160 mmHg or an average DBP ≥100 mmHg
* Known severe renal impairment
* High risk Proliferative Diabetic Retinopathy
* History of retinal disease in the study eye other than diabetic retinopathy
* History of retinal detachment (with or without repair) in the study eye
* History of vitrectomy, trabeculectomy, or other filtration surgery in the study eye
* Any prior focal or grid laser photocoagulation or any prior PRP in the study eye
* Current or planned pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2023-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: INFINITY Medical Monitor, MD, Study Chair — Adverum Biotechnologies, Inc.
Locations (14):
- United States (13):
  - Adverum Clinical Site, Phoenix, Arizona
  - Adverum Clinical Site, Bakersfield, California
  - Adverum Clinical Site, Beverly Hills, California
  - Adverum Clinical Site, Golden, Colorado
  - Adverum Clinical Site, Deerfield Beach, Florida
  - Adverum Clinical Site, Reno, Nevada
  - Adverum Clinical Site, Philadelphia, Pennsylvania
  - Adverum Clinical Site, West Columbia, South Carolina
  - Adverum Clinical Site, Nashville, Tennessee
  - Adverum Clinical Site, Abilene, Texas
  - Adverum Clinical Site, Austin, Texas
  - Adverum Clinical Site, Houston, Texas
  - Adverum Clinical Site, The Woodlands, Texas
- Adverum Clinical Site, Arecibo, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two doses of ADVM-022 (Ixo-vec) were investigated, administered with or without a prior loading dose of Aflibercept. The control group received the initial loading dose of Aflibercept (Day 1) but received a Sham injection on Day 8 instead of Ixo-vec. Only one eye was selected as the study eye. After the assigned intravitreal (IVT) injections on Days 1 and 8, clinic visits were on Weeks 2, 4, and every 4 weeks up to Week 96. Consenting participants then entered a long-term follow-up study.
Pre-assignment Details: Participants with initial diagnosis of DME within 6 months of screening, and who had received up to 2 prior injections of anti-VEGF therapy in the study eye (0, 1 or 2) were eligible for enrollment. If a prior anti-VEGF had been administered to the study eye, in the judgement of the Investigator, there must have been a meaningful CST response (e.g., ≥ 10% reduction) and no adverse reaction to the anti-VEGF (e.g., intraocular inflammation).
Groups:
- ADVM-022 6E11 vg/Eye: 6E11 vg/eye ADVM-022 +/- aflibercept 2mg IVT
  6E11 vg/eye of ADVM-022: ADVM-022 (AAV.7m8-aflibercept) is a recombinant, replication-incompetent adeno-associated virus (AAV.7m8) gene therapy vector carrying a coding sequence for aflibercept
  Aflibercept: Commercially available Active Comparator
- ADVM-022 2E11 vg/Eye: 2E11 vg/eye ADVM-022 +/- aflibercept 2mg IVT
  2E11 vg/eye of ADVM-022: ADVM-022 (AAV.7m8-aflibercept) is a recombinant, replication-incompetent adeno-associated virus (AAV.7m8) gene therapy vector carrying a coding sequence for aflibercept
  Aflibercept: Commercially available Active Comparator
- Aflibercept + Sham: Aflibercept 2mg IVT
  Aflibercept: Commercially available Active Comparator
Period: Overall Study
Arm/Group | ADVM-022 6E11 vg/Eye | ADVM-022 2E11 vg/Eye | Aflibercept + Sham
Started | 13 | 13 | 10
Modified ITT (mITT) Population (The modified ITT (mITT) population included all randomized participants who received study treatment at both Day 1 (Aflibercept or Sham) and Day 8 (ADVM-022 or Sham). Two participants (1 randomized to ADVM-022-6E11 vg/Eye and 1 randomized to Aflibercept + Sham) treated on Day 1 were withdrawn by the Sponsor prior to Day 8 due to the syringe manufacturer warning letter (in the UK) advising against intra-ocular use. These two participants are not included in mITT. They reported no adverse events.) | 12 | 13 | 9
Completed | 12 | 9 | 7
Not Completed | 1 | 4 | 3
Not completed — Death | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 2 | 2
Not completed — Subject Discontinued by the Sponsor | 1 | 0 | 1
Not completed — Pre-existing medical condition | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: ITT (Intent to Treat) Population included all participants randomized to treatment. Participants were analyzed as randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | ADVM-022 6E11 vg/Eye | ADVM-022 2E11 vg/Eye | Aflibercept + Sham | Total
Number analyzed (Participants) | 13 | 13 | 10 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.8 (5.94) | 60.5 (8.28) | 56.6 (5.68) | 60.3 (7.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 5 | 15
  Male | 7 | 9 | 5 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 6 | 20
  Not Hispanic or Latino | 6 | 6 | 4 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 0 | 4
  White | 11 | 10 | 10 | 31
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Worsening of DME Disease Activity in the Study Eye.
Description: Time to worsening of DME disease activity in the study eye through 96 weeks.
  Time to worsening of DME disease activity defined by either: An increase in CST > 50 µm as assessed by SD-OCT compared to the lower of the two CST measurements recorded at Day 1 or Week 4; A loss of > 5 letters in BCVA due to worsening DME disease activity compared to the higher of the two BCVA measurements recorded at Day 1 or Week 4. Number of weeks was relative to Day 1.
Time Frame: Day 1 through 96 weeks
Population: The Modified Intent to Treat population (mITT) was analyzed for this endpoint (mITT population includes all randomized participants who received study treatment at both Day 1 [Aflibercept or Sham] and Day 8 [Ixo-vec or Sham]).
Measure: Median (90% Confidence Interval); unit: Weeks
Units Other Than Participants: Study Eyes
Arm/Group | ADVM-022 6E11 vg/Eye | ADVM-022 2E11 vg/Eye | Aflibercept + Sham
Number analyzed (Participants) | 12 | 13 | 9
Number analyzed (Study Eyes) | 12 | 13 | 9
Weeks | 82.1 [12.1 to NA] — The upper limit of the 90% confidence interval was not calculable because an insufficient number of participants experienced the event by the final time point for assessment. | 96.1 [20.6 to NA] — The upper limit of the 90% confidence interval was not calculable because an insufficient number of participants experienced the event by the final time point for assessment. | 19.1 [12.7 to 24.0]

2. Secondary Outcome: Incidence of Ocular Adverse Events (AEs)
Description: Incidence of ocular adverse events (AEs) through 96 weeks
Time Frame: 96 weeks
Population: mITT population: participants who received treatment on Day 1 (aflibercept or Sham) and Day 8 (Ixo-vec or Sham) analyzed based on treatments they received on Days 1 and 8. Ocular adverse events are presented for the Study Eye only.
  Note: two participants who were discontinued prior to Day 8 are not included in the mITT population. These two participants reported no adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | ADVM-022 6E11 vg/Eye | ADVM-022 2E11 vg/Eye | Aflibercept + Sham
Number analyzed (Participants) | 12 | 13 | 9
Participants | 12 | 13 | 9

3. Secondary Outcome: Incidence of Non-ocular Adverse Events (AEs)
Description: Incidence of non-ocular adverse events (AEs) through 96 weeks.
Time Frame: Day 1 through 96 weeks
Population: mITT population: participants who received treatment on Day 1 (aflibercept or Sham) and Day 8 (Ixo-vec or Sham) analyzed based on treatments they received on Days 1 and 8.
  Note: two participants who were discontinued prior to Day 8 are not included in the mITT population. These two participants reported no adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | ADVM-022 6E11 vg/Eye | ADVM-022 2E11 vg/Eye | Aflibercept + Sham
Number analyzed (Participants) | 12 | 13 | 9
Participants | 9 | 9 | 7

4. Secondary Outcome: Change From Baseline Central Subfield Thickness (CST) in Study Eye
Description: Central subfield thickness is a measurement of the thickness of the retina in a circular area around the fovea. Least squares mean change from Baseline in central subfield thickness at Week 96 is presented for the study eye.
Time Frame: Baseline through 96 weeks
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: micrometers
Units Other Than Participants: Study Eyes
Arm/Group | ADVM-022 6E11 vg/Eye | ADVM-022 2E11 vg/Eye | Aflibercept + Sham
Number analyzed (Participants) | 12 | 13 | 9
Number analyzed (Study Eyes) | 12 | 13 | 9
micrometers | -84.4 [-124.0 to -44.9] | -129.7 [-172.2 to -87.3] | -129.7 [-176.9 to -82.4]

5. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) Score Over Time in the Study Eye
Description: Least squares mean change from Baseline in BCVA score over time was measured over time through week 96 in the study eye by ETDRS letters.
Time Frame: 96 weeks
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: ETDRS letters
Units Other Than Participants: Study Eyes
Groups:
- ADVM-022 6E11vg/Eye: 6E11 vg/eye ADVM-022 +/- aflibercept 2mg IVT
  6E11 vg/eye of ADVM-022: ADVM-022 (AAV.7m8-aflibercept) is a recombinant, replication-incompetent adeno-associated virus (AAV.7m8) gene therapy vector carrying a coding sequence for aflibercept
  Aflibercept: Commercially available Active Comparator
Arm/Group | ADVM-022 6E11vg/Eye | ADVM-022 2E11 vg/Eye | Aflibercept + Sham
Number analyzed (Participants) | 12 | 13 | 9
Number analyzed (Study Eyes) | 12 | 13 | 9
ETDRS letters | -11.9 [-20.7 to -3.2] | 10.1 [0.4 to 19.8] | 17.1 [7.1 to 27.0]

6. Secondary Outcome: Frequency of Supplemental Aflibercept Injections (2 mg IVT) in the Study Eye Over Time During the Study
Description: Frequency of supplemental aflibercept (2 mg IVT) injections was assessed in the study eye over time during the study.
  Participants were analyzed according to the study treatments they actually received on Days 1 and 8.
  The rate of supplemental aflibercept per year = Total number of supplemental aflibercept injections / Total years at-risk (at-risk duration starting at Day 8).
Time Frame: Day 1 through 96 weeks
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: Injections/year
Units Other Than Participants: Study Eyes
Arm/Group | ADVM-022 6E11 vg/Eye | ADVM-022 2E11 vg/Eye | Aflibercept + Sham
Number analyzed (Participants) | 12 | 13 | 9
Number analyzed (Study Eyes) | 12 | 13 | 9
Injections/year | 1.001 [0.022 to 1.979] | 0.423 [0.055 to 0.792] | 5.54 [3.058 to 8.029]

7. Secondary Outcome: Incidence of 2-step Improvement in Diabetic Retinopathy Severity Score (DRSS) in the Study Eye Over Time
Description: Diabetic Retinopathy Severity Score was determined by the Central Reading Center using ultra-wide field color retinopathy fundus photography. The score represents a comprehensive evaluation of retinal health, including the presence of microaneurysms, hemorrhages, and other abnormalities in the retina of the study eye. The score ranges from 10 to 85 and is divided into 13-steps used to classify increasing diabetic retinopathy severity (with higher scored indicating more advanced stages of Diabetic Retinopathy). In this endpoint a 2-step improvement indicates an improvement in a participant across 2 steps of the 13-step scale.
Time Frame: From Day 1 through 96 weeks
Population: The Modified Intent to Treat population (mITT) was analyzed for this endpoint (mITT population includes all randomized participants treated on both Day 1 [Aflibercept or Sham] and Day 8 [Ixo-vec or Sham]). Only mITT participants whose Baseline Score permitted a ≥ 2 step DRSS improvement were eligible for this analysis. The incidence of 2-step improvement in DRSS score over time at Week 96 is presented.
Measure: Count of Participants; unit: Participants
Arm/Group | ADVM-022 6E11 vg/Eye | ADVM-022 2E11 vg/Eye | Aflibercept + Sham
Number analyzed (Participants) | 11 | 11 | 8
Participants | 8 | 8 | 4

8. Secondary Outcome: Incidence of 3-step Improvement in DRSS (Diabetic Retinopathy Severity Score) in the Study Eye Over Time
Description: Diabetic Retinopathy Severity Score was determined by the Central Reading Center using ultra-wide field color retinopathy fundus photography. The score represents a comprehensive evaluation of retinal health, including the presence of microaneurysms, hemorrhages, and other abnormalities in the retina of the study eye. The score ranges from 10 to 85 and is divided into 13-steps used to classify increasing diabetic retinopathy severity (with higher scored indicating more advanced stages of Diabetic Retinopathy). In this endpoint a 3-step improvement indicates an improvement in a participant across 3 steps of the 13-step scale.
Time Frame: From Day 1 through 96 weeks
Population: The Modified Intent to Treat population (mITT) was analyzed for this endpoint (mITT population includes all randomized participants treated on both Day 1 [Aflibercept or Sham] and Day 8 [Ixo-vec or Sham]). Only mITT participants whose Baseline Score permitted a ≥3 step DRSS improvement were eligible for this analysis. The incidence of 3-step improvement in DRSS score over time at Week 96 is presented. Visits with a 3-step or greater improvement in DRSS were considered separate events.
Measure: Count of Participants; unit: Participants
Arm/Group | ADVM-022 6E11 vg/Eye | ADVM-022 2E11 vg/Eye | Aflibercept + Sham
Number analyzed (Participants) | 8 | 8 | 5
Participants | 3 | 4 | 0

9. Secondary Outcome: Incidence of 2-step Worsening in DRSS (Diabetic Retinopathy Severity Score) in the Study Eye Over Time
Description: Diabetic Retinopathy Severity Score was determined by the Central Reading Center using ultra-wide field color retinopathy fundus photography. The score represents a comprehensive evaluation of retinal health, including the presence of microaneurysms, hemorrhages, and other abnormalities in the retina of the study eye. The score ranges from 10 to 85 and is divided into 13-steps used to classify increasing diabetic retinopathy severity (with higher scored indicating more advanced stages of Diabetic Retinopathy). In this endpoint a 2-step worsening indicates a worsening across 2 steps of the 13-step scale.
  Note: 2-step worsening in DRSS was observed in 2 participants in both the control arm and the ADVM-022 6E11 vg/eye arm. These participants experienced ocular adverse events which may have contributed, at least in part, to the worsening in DRSS. This included one participant in the ADVM-022 6E11 vg/eye arm who had a SUSAR of Hypotony of eye (secondary to intraocular inflammation).
Time Frame: From Day 1 through 96 weeks
Population: The Modified Intent to Treat population (mITT) was analyzed for this endpoint (mITT population includes all randomized participants who received study treatment at both Day 1 [Aflibercept or Sham] and Day 8 [Ixo-vec or Sham]). The incidence of 2-step worsening in DRSS score over time at Week 96 is presented. Visits with a 2-step or greater worsening in DRSS were considered separate events.
Measure: Count of Participants; unit: Participants
Arm/Group | ADVM-022 6E11 vg/Eye | ADVM-022 2E11 vg/Eye | Aflibercept + Sham
Number analyzed (Participants) | 12 | 13 | 9
Participants | 2 | 0 | 2

10. Secondary Outcome: Incidence of 3-step Worsening in DRSS (Diabetic Retinopathy Severity Score) in the Study Eye Over Time
Description: Diabetic Retinopathy Severity Score was determined by the Central Reading Center using ultra-wide field color retinopathy fundus photography. The score represents a comprehensive evaluation of retinal health, including the presence of microaneurysms, hemorrhages, and other abnormalities in the retina of the study eye. The score ranges from 10 to 85 with higher scored indicating more advanced stages of Diabetic Retinopathy. The incidence of 3-step worsening in DRSS score over time at Week 96 is presented. Visits with a 3-step or greater worsening in DRSS were considered separate events.
  Note: 3-step worsening in DRSS was observed in one participant each in the control arm and the ADVM-022 6E11 vg/eye arm. Both participants experienced ocular adverse events which may have contributed, at least in part, to the worsening in DRSS. This included one participant in the ADVM-022 6E11 vg/eye arm who had a SUSAR of Hypotony of eye (secondary to intraocular inflammation).
Time Frame: From Day 1 through 96 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ADVM-022 6E11 vg/Eye | ADVM-022 2E11 vg/Eye | Aflibercept + Sham
Number analyzed (Participants) | 12 | 13 | 9
Participants | 1 | 0 | 1

11. Secondary Outcome: Occurrence of Any Vision Threatening Complications in the Study Eye (Anterior Segment Neovascularization, Vitreous Hemorrhage, or Any Other High-risk Proliferative DR, or Tractional Retinal Detachment) Over Time Through Week 96
Description: Occurrence of any vision threatening complication over time though 96 weeks. Results present the incidence of participants who experienced "Any Vision Threatening Complications" (defined as any Vitreous Haemorrhage adverse event (AE), Anterior Segment Neovascularization AE, High-risk proliferative DR (defined as DSSR >= 71), or Tractional Retinal Detachment AE) in the study eye from Day 1 through 96 weeks.
  Note: AEs of Vitreous Haemorrhage and High-risk proliferative DR were reported in 1 participant in the control arm and in 2 separate participants in the 6E11 vg/eye arm. No AE of Tractional Retinal Detachment or Anterior Segment Neovascularization occurred.
Time Frame: From Day 1 through 96 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ADVM-022 6E11 vg/Eye | ADVM-022 2E11 vg/Eye | Aflibercept + Sham
Number analyzed (Participants) | 12 | 13 | 9
Participants | 2 | 0 | 1

12. Secondary Outcome: Incidence of CST <300 μm Over Time Through Week 96 in the Study Eye
Description: Central subfield thickness is a measurement of the thickness of the retina in a circular area around the fovea. Incidence of participants with Central subfield thickness of less than 300 μm over time in the study eye through Week 96 is presented.
Time Frame: Day 1 through 96 weeks
Population: The Modified Intent to Treat population (mITT) was analyzed for this endpoint (mITT population includes all randomized participants who received study treatment at both Day 1 [Aflibercept or Sham] and Day 8 [Ixo-vec or Sham]). Incidence through last visit represent the last visit through Week 96 with non-missing CST data.
Measure: Count of Participants; unit: Participants
Arm/Group | ADVM-022 6E11 vg/Eye | ADVM-022 2E11 vg/Eye | Aflibercept + Sham
Number analyzed (Participants) | 12 | 13 | 9
Participants | 8 | 6 | 4

ADVERSE EVENTS:
Time Frame: Adverse event data are presented from study treatment on Day 1 through Week 96.
Description: The modified Intent to Treat (mITT) Population was analyzed - included all participants who received treatment on Day 1 (Aflibercept or Sham) and Day 8 (Ixo-vec or Sham) and data summarized based on treatments participants received on Days 1 and 8. The mITT population does not include 2 participants who were discontinued prior to Day 8. Neither of these participants reported any adverse events. Ocular adverse events are presented for the Study Eye only (no SAEs were reported in the fellow eye).
Arm/Group | ADVM-022 6E11 vg/Eye | ADVM-022 2E11 vg/Eye | Aflibercept + Sham
All-Cause Mortality (participants affected / at risk) | 0/12 | 1/13 | 0/9
Serious Adverse Events (participants affected / at risk) | 9/12 | 8/13 | 4/9
Other Adverse Events (participants affected / at risk) | 12/12 | 13/13 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ADVM-022 6E11 vg/Eye (N=12) | ADVM-022 2E11 vg/Eye (N=13) | Aflibercept + Sham (N=9)
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 4 | 2 | 1 — Ocular SAEs are presented for the Study Eye only.
Cataract subcapsular (Eye disorders) | 2 | 3 | 0 — Ocular SAEs are presented for the Study Eye only.
Visual impairment (Eye disorders) | 4 | 0 | 0 — Ocular SAEs are presented for the Study Eye only.
Hypotony of eye (Eye disorders) | 3 | 0 | 0 — Ocular SAEs are presented for the Study Eye only.
Iridocyclitis (Eye disorders) | 2 | 0 | 0 — Ocular SAEs are presented for the Study Eye only.
Angle closure glaucoma (Eye disorders) | 1 | 0 | 0 — Ocular SAEs are presented for the Study Eye only.
Cataract nuclear (Eye disorders) | 0 | 1 | 0 — Ocular SAEs are presented for the Study Eye only.
Choroidal effusion (Eye disorders) | 1 | 0 | 0 — Ocular SAEs are presented for the Study Eye only.
Cystoid macular oedema (Eye disorders) | 0 | 0 | 1 — Ocular SAEs are presented for the Study Eye only.
Vitritis (Eye disorders) | 1 | 0 | 0 — Ocular SAEs are presented for the Study Eye only.
Diabetic gastroparesis (Gastrointestinal disorders) | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0 | 0
Gangrene (Infections and infestations) | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1
Osteomyelitis acute (Infections and infestations) | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Carotid artery occlusion (Nervous system disorders) | 1 | 0 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 2 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Hypertensive emergency (Vascular disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
Peripheral artery occlusion (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ADVM-022 6E11 vg/Eye (N=12) | ADVM-022 2E11 vg/Eye (N=13) | Aflibercept + Sham (N=9)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1 | 0
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0 | 1
Iridocyclitis (Eye disorders) | 7 | 6 | 0 — Ocular AEs are presented for the Study Eye only.
Anterior chamber cell (Eye disorders) | 6 | 4 | 3 — Ocular AEs are presented for the Study Eye only.
Iris transillumination defect (Eye disorders) | 8 | 4 | 0 — Ocular AEs are presented for the Study Eye only.
Iris adhesions (Eye disorders) | 6 | 5 | 0 — Ocular AEs are presented for the Study Eye only.
Ocular hypertension (Eye disorders) | 3 | 3 | 4 — Ocular AEs are presented for the Study Eye only.
Conjunctival haemorrhage (Eye disorders) | 5 | 3 | 2 — Ocular AEs are presented for the Study Eye only.
Diabetic retinal oedema (Eye disorders) | 4 | 3 | 3 — Ocular AEs are presented for the Study Eye only.
Pigment dispersion syndrome (Eye disorders) | 3 | 3 | 0 — Ocular AEs are presented for the Study Eye only.
Cataract (Eye disorders) | 4 | 2 | 0 — Ocular AEs are presented for the Study Eye only.
Keratic precipitates (Eye disorders) | 2 | 3 | 0 — Ocular AEs are presented for the Study Eye only.
Vitreous floaters (Eye disorders) | 4 | 1 | 0 — Ocular AEs are presented for the Study Eye only.
Cataract subcapsular (Eye disorders) | 4 | 1 | 0 — Ocular AEs are presented for the Study Eye only.
Iris hyperpigmentation (Eye disorders) | 2 | 3 | 0 — Ocular AEs are presented for the Study Eye only.
Iritis (Eye disorders) | 2 | 3 | 0 — Ocular AEs are presented for the Study Eye only.
Uveitis (Eye disorders) | 3 | 2 | 0 — Ocular AEs are presented for the Study Eye only.
Decrease in intraocular pressure (Eye disorders) | 3 | 1 | 0 — Ocular AEs are presented for the Study Eye only.
Corneal striae (Eye disorders) | 3 | 1 | 0 — Ocular AEs are presented for the Study Eye only.
Punctate keratitis (Eye disorders) | 3 | 1 | 0 — Ocular AEs are presented for the Study Eye only.
Anterior chamber flare (Eye disorders) | 2 | 0 | 1 — Ocular AEs are presented for the Study Eye only.
Lenticular pigmentation (Eye disorders) | 1 | 2 | 0 — Ocular AEs are presented for the Study Eye only.
Vitreous detachment (Eye disorders) | 2 | 1 | 0 — Ocular AEs are presented for the Study Eye only.
Corneal oedema (Eye disorders) | 2 | 0 | 0 — Ocular AEs are presented for the Study Eye only.
Flat anterior chamber of eye (Eye disorders) | 2 | 0 | 0 — Ocular AEs are presented for the Study Eye only.
Iris atrophy (Eye disorders) | 2 | 0 | 0 — Ocular AEs are presented for the Study Eye only.
Mydriasis (Eye disorders) | 1 | 1 | 0 — Ocular AEs are presented for the Study Eye only.
Posterior capsule opacification (Eye disorders) | 2 | 0 | 0 — Ocular AEs are presented for the Study Eye only.
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 1 — Ocular AEs are presented for the Study Eye only.
Vitreous opacities (Eye disorders) | 1 | 1 | 0 — Ocular AEs are presented for the Study Eye only.
Ocular hypotension (Eye disorders) | 1 | 0 | 0 — Ocular AEs are presented for the Study Eye only.
Vision blurred (Eye disorders) | 0 | 0 | 1 — Ocular AEs are presented for the Study Eye only.
Cataract nuclear (Eye disorders) | 1 | 0 | 0 — Ocular AEs are presented for the Study Eye only.
Chalazion (Eye disorders) | 1 | 0 | 0 — Ocular AEs are presented for the Study Eye only.
Ciliary body disorder (Eye disorders) | 1 | 0 | 0 — Ocular AEs are presented for the Study Eye only.
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 0 — Ocular AEs are presented for the Study Eye only.
Corneal erosion (Eye disorders) | 1 | 0 | 0 — Ocular AEs are presented for the Study Eye only.
Diabetic retinopathy (Eye disorders) | 1 | 0 | 0 — Ocular AEs are presented for the Study Eye only.
Epiretinal membrane (Eye disorders) | 0 | 1 | 0 — Ocular AEs are presented for the Study Eye only.
Eyelid margin crusting (Eye disorders) | 1 | 0 | 0 — Ocular AEs are presented for the Study Eye only.
Eyelid ptosis (Eye disorders) | 0 | 1 | 0 — Ocular AEs are presented for the Study Eye only.
Foreign body sensation in eyes (Eye disorders) | 0 | 1 | 0 — Ocular AEs are presented for the Study Eye only.
Hypotony (Eye disorders) | 1 | 0 | 0 — Ocular AEs are presented for the Study Eye only.
Hypotony maculopathy (Eye disorders) | 1 | 0 | 0 — Ocular AEs are presented for the Study Eye only.
IOP 5mmHG Post injection (Eye disorders) | 0 | 0 | 1 — Ocular AEs are presented for the Study Eye only.
Narrow anterior chamber angle (Eye disorders) | 0 | 0 | 1 — Ocular AEs are presented for the Study Eye only.
Ocular discomfort (Eye disorders) | 1 | 0 | 0 — Ocular AEs are presented for the Study Eye only.
Periorbital oedema (Eye disorders) | 1 | 0 | 0 — Ocular AEs are presented for the Study Eye only.
Periorbital pain (Eye disorders) | 1 | 0 | 0 — Ocular AEs are presented for the Study Eye only.
Photophobia (Eye disorders) | 0 | 1 | 0 — Ocular AEs are presented for the Study Eye only.
Swelling of eyelid (Eye disorders) | 1 | 0 | 0 — Ocular AEs are presented for the Study Eye only.
Visual impairment (Eye disorders) | 0 | 1 | 0 — Ocular AEs are presented for the Study Eye only.
Vitreal cells (Eye disorders) | 0 | 1 | 0 — Ocular AEs are presented for the Study Eye only.
Vitreoretinal traction syndrome (Eye disorders) | 1 | 0 | 0 — Ocular AEs are presented for the Study Eye only.
Vitreous haze (Eye disorders) | 1 | 0 | 0 — Ocular AEs are presented for the Study Eye only.
Toothache (Gastrointestinal disorders) | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Gallbladder polyp (Hepatobiliary disorders) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 3 | 0 | 3
Urinary tract infection (Infections and infestations) | 2 | 0 | 1
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0
Eye infection (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection staphylococcal (Infections and infestations) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 2
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hyphaema (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Intraocular pressure increased (Investigations) | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 4 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Degenerative bone disease (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 2 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 1
Cerebral ventricle dilatation (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0
Device dislocation (Product Issues) | 1 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Renal atrophy (Renal and urinary disorders) | 0 | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0 | 0
Pelvic fluid collection (Reproductive system and breast disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 3
Aortic arteriosclerosis (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0
Gastrooesophageal hypot disease (Gastrointestinal disorders) | 0 | 2 | 0

LIMITATIONS AND CAVEATS:
Although this study was initiated as a randomized, double-masked study, the Sponsor and the independent data monitoring committee agreed to unmask the study following an ocular suspected unexpected serious adverse reaction (SUSAR) of Hypotony and concerns regarding the appropriate management of ocular inflammation and hypotony. All participants had reached the 12-week assessment at the time of unmasking.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to postponement of single-site study publications until after publication of all multi-center study results, until notification by the Sponsor that a multi-center publication is not planned, or until eighteen (18) months after final database lock.

DOCUMENTS (2):
  • Study Protocol (2021-08-05): https://cdn.clinicaltrials.gov/large-docs/27/NCT04418427/Prot_002.pdf
  • Statistical Analysis Plan (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/27/NCT04418427/SAP_003.pdf